CLINICAL TRIAL: NCT03950635
Title: Controlled Dietary Interventions in Patients with Melanoma
Brief Title: Dietary Intervention in Patients with a History of Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively Complete
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0857; NCI-2019-02496 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0857 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-05-06; First posted 2019-05-15 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (fiber-rich diet) (Experimental): Patients consume a whole-foods, fiber-rich diet for 6 weeks.
  Interventions: Dietary Supplement: Dietary Intervention; Other: Questionnaire Administration
- Group II (ketogenic diet) (Experimental): Patients consume a high fat, low carbohydrate (ketogenic) diet for 6 weeks.
  Interventions: Dietary Supplement: Dietary Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Dietary Supplement: Dietary Intervention — Consume whole-foods, fiber-rich diet
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
  Arms: Group I (fiber-rich diet)
Dietary Supplement: Dietary Intervention — Consume high fat, low carbohydrate (ketogenic) diet
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
  Arms: Group II (ketogenic diet)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This research trial studies the effects of diet in patients with a history of melanoma. We are studying the impact of 2 different diets; a whole-foods, fiber-rich diet and a ketogenic diet. Participants will be assigned to one of these diets. During this study, participants will be provided all food at no cost for the entire 6-week study. Food can be picked up or shipped to the participant's home. However, participants will need to come into MD Anderson Cancer Center in Houston, TX, for the initial screening visit and for blood tests every 2 weeks during the study.

DETAILED DESCRIPTION:
Study Background:

Whole-foods, fiber-rich diet rationale: Recent studies have shown that the gut microbiome (the trillions of bacteria that live in our intestines) can influence our immune system function. Diet plays a key role in shaping the gut microbiome. We will examine the effects of a whole-food, fiber-rich diet on the gut microbiome within patients with a history of melanoma.

Ketogenic diet rationale: The ketogenic diet is a very-low-carbohydrate, high-fat diet. The goal of this diet is to change the body's fuel source from carbohydrates to fat and to lower levels of insulin. We will examine the effects of a ketogenic diet to change metabolism within patients with a history of melanoma.

Who can participate?

To be eligible for the study, participants must meet the following criteria:

* Be at least 18 years old;
* Meet the study requirements for Body Mass Index (BMI);
* Have had melanoma within the last 5 years;
* Be cancer-free at the start of the trial;
* Have not received systemic therapy within the last year; and
* Have no medical issues that would make them unable to follow these eating plans.

Study Design:

Our study will enroll up to 10 participants to each diet (high-fiber or ketogenic). After screening, participants will have baseline assessment performed that will include collecting diet information, blood and fecal samples, and body composition information. Participants will then eat the provided diets for the next 6 weeks while coming in every 2 weeks for blood and stool specimen collection. Six (6)weeks after the diet intervention is complete, participants will come back to MD Anderson for one last end of study visit.

Who makes the meals?:

All calorie-containing food and beverages will be provided by either the MD Anderson Cancer Center Bionutrition Research Core or Savor Health (a third-party vendor contracted by MD Anderson).

Costs: There will be no cost to participate in this study.

Benefits:

All food and beverages you will eat as part of this study will be provided by the study and can be shipped directly to your home. The results will be used to help us design future dietary intervention trials in Melanoma patients receiving immunotherapy. Please note, participants can withdraw from the study at any time without consequences.

Study PI: Dr. Jennifer McQuade

NCT#: NCT03950635

Contact Info:

Melanoma Medical Oncology (713)-792-5500 MelanomaDiet@mdanderson.org

Where: MD Anderson Cancer Center, Department of Melanoma Medical Oncology, Houston, TX

ELIGIBILITY:
Inclusion Criteria:

* Melanoma resected within the last 5 years, currently no evidence of disease (NED) and not on systemic therapy.
* Body mass index (BMI) 18.5-40 kg/m^2.
* English-speaking.
* Self-reported willingness to exclusively eat the provided diets.
* Self-reported willingness to comply with scheduled visits, undergo venipuncture, provide stool samples.
* Creatinine (Cr) < 1.5 mg/dL.
* Liver function tests (LFTs) 2 x upper limit of normal (ULN).
* Fasting glucose < 125 mg/dL.
* Women of child-bearing (WOCP) potential must have negative urine pregnancy test (UPT) within 1 week prior to dual x-ray absorptiometry (DEXA) scan.

Exclusion Criteria:

* Systemic treatment for melanoma within the past 1 year.
* Medical contraindications to the intervention diet as determined by the treating physician.
* Self-reported major dietary restrictions related to the intervention.
* Diagnosis of diabetes mellitus type I or type II that requires medical treatment.
* Unable or unwilling to undergo study procedures.
* Antibiotic use within the last 30 days (self-reported and/or noted by the treating physician).
* Regularly taking probiotics, fiber supplements, or bile acid sequestrants, exogenous ketones, weight loss supplements, appetite suppressants, carnitine supplements, creatine supplements or diuretics within the last 30 days (self-reported and/or noted by the treating physician).
* Currently following a ketogenic diet with > 70% calories derived from fat or consuming > 40 grams of fiber per day or a vegetarian or vegan diet.
* Current self-reported smoker or heavy drinker (defined as > 14 drinks per week) or current self-reported illicit drug use.
* Pregnant or lactating.
* Low density lipoprotein (LDL) > 200 mg/dL (within 28 days of screening).
* Triglycerides > 350 mg/dL (within 28 days of screening).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Feasibility of conducting a controlled feeding study in melanoma patients | Up to 1 year
  Defined by >= 25% of eligible patients enrolling on the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer McQuade, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org
- See also: https://www.mdanderson.org/patients-family/diagnosis-treatment/clinical-trials/clinical-trials-index/clinical-trials-detail.ID2018-0857.html — http://www.mdanderson.org